CLINICAL TRIAL: NCT05379855
Title: The Effects of Atropine Eyedrops on Ocular Alignment and Binocular Vision
Brief Title: A-eyedrops on Ocular Alignment and Binocular Vision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Chen Zhao, Vice President of Department of Ophthalmology and Visual Science, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022C-PEDIG-Atropine
Record Dates: First submitted 2022-04-24; First posted 2022-05-18 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Exotropia; Exophoria; Myopia
Keywords: atropine; myopia; ocular alignment; binocular vision; exotropia; exophoria
MeSH Terms: conditions — Exotropia; Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.05% atropine group (Experimental): Subjects received 0.05% atropine eye drops (0.1% sodium hyaluronate as a solution) both eyes once every night. Eye drops are prepackaged with identical eye drops bottle, pasted with number and shelf life, and stored in 4℃.
  Interventions: Drug: 0.05% atropine eye drops
- placebo group (Placebo Comparator): Subjects of the control group received placebo eye drops (0.1% sodium hyaluronate ophthalmic solution) both eyes once every night. Eye drops are prepackaged with identical eye drops bottle, pasted with number and shelf life, and stored in 4℃.
  Interventions: Drug: placebo eye drops (0.1% sodium hyaluronate ophthalmic solution)
- 0.01% atropine group (Experimental): Subjects received 0.01% atropine eye drops (0.1% sodium hyaluronate as a solution) both eyes once every night. Eye drops are prepackaged with identical eye drops bottle, pasted with number and shelf life, and stored in 4℃.
  Interventions: Drug: 0.01% atropine eye drops

INTERVENTIONS:
Drug: 0.01% atropine eye drops — using 0.01% atropine eye drops for both eyes every night
  Arms: 0.01% atropine group
Drug: placebo eye drops (0.1% sodium hyaluronate ophthalmic solution) — using placebo eye drops (0.1% sodium hyaluronate ophthalmic solution) for both eyes every night
  Arms: placebo group
Drug: 0.05% atropine eye drops — using 0.05% atropine eye drops for both eyes every night
  Arms: 0.05% atropine group

SUMMARY:
Atropine is a non-selective muscarinic acetylcholine (M) receptor antagonist that paralyzes the ciliary muscle, dilates the pupil, and reduces the power of accommodation. Current studies have confirmed the effect of low concentrations of atropine drops in slowing the progression of myopia. In the atropine treatment for myopia (ATOM2) study, there was a rapid and dose-dependent decrease in accommodation after atropine drops: after 2 weeks of use, accommodation decreased from baseline 16.2D to 11.3D (4.9D) in the 0.01% atropine drops group, from baseline 16.7D to 3.8D (12.9D) in the 0.1% atropine group, and from baseline 15.8 D to 2.2 D (13.6 D) in the 0.5% atropine group; one year after withdrawal, there was some recovery of the accommodation in all the three groups, but it was still lower than the baseline values for each group, with a mean decrease of 2.56 D.Similar results were found in the Low-concentration Atropine for Myopia Progression (LAMP) Study by Janson C. Yam, 0.05% atropine drops reduced the accommodation by approximately 2D on average after 1 year of treatment.

In general, if accommodation decreases by 2D or more compared to normal values, accommodation insufficiency is considered. There is a linkage between accommodation and convergence called accommodative convergence-to-accommodation (AC/A) which is closely related to exotropia. It was reported that the amount of accommodation required to maintain binocular fusion in patients with intermittent exotropia was greater than that of normal controls. In addition, pupil size and visual acuity are also factors that affect accommodation. In summary, the reduced accommodation amplitude, pupil dilation, and blurred near vision caused by atropine drops would affect the progression of intermittent exotropia and the ocular alignment after the surgery. In most cases, the reduced accommodation and convergence might induce exotropia, but in some patients, they may use more accommodative stimuli to compensate the insufficiency of accommodation, and there may be an increase in convergence or even esotropia.

Taken together, due to the effect of atropine drops on pupil size, near visual acuity, and accommodation amplitude, the investigators hypothesize that atropine drops are likely to affect binocular vision and ocular alignment in patients with exotropia and exophoria.

DETAILED DESCRIPTION:
The prevalence of myopia in the world has exceeded 25% and is increasing year by year. Asia, especially China, is an area with high incidence of myopia. It is reported that the prevalence of myopia in children and adolescents in China was 53.6% in 2018. Low concentration atropine eye drops is one of the effective means to slow the progression of myopia. At present, low concentration atropine eye drops have been widely used in China, but its long-term efficacy and possible side effects still need to be studied.

Atropine is a non-selective muscarinic acetylcholine (M) receptor antagonist that paralyzes the ciliary muscle, dilates the pupil, and reduces the power of accommodation. Current studies have confirmed the effect of low concentrations of atropine drops in slowing the progression of myopia. In the ATOM2 study, there was a rapid and dose-dependent decrease in accommodation after atropine drops: after 2 weeks of use, accommodation decreased from baseline 16.2D to 11.3D (4.9D) in the 0.01% atropine drops group, from baseline 16.7D to 3.8D (12.9D) in the 0.1% atropine group, and from baseline 15.8 D to 2.2 D (13.6 D) in the 0.5% atropine group; after 1 year of discontinuation, there was some recovery of the accommodation in all the three groups, but it was still lower than the baseline values for each group, with a mean decrease of 2.56 D. Similar results were found in the LAMP study by Janson C. Yam, 0.05% atropine drops reduced the accommodation by approximately 2D on average after 1 year of treatment. In general, if accommodation decreases by 2D or more compared to normal values, accommodation insufficiency is considered. There is a linkage between accommodation and convergence, therefore the decrease of accommodation will also affect the binocular vision. Above all, the effect of atropine eye drops on pupil size, near visual acuity, amplitude of accommodation which is still impaired after 1 years' withdrawal, make us have many concerns and doubts about indications of atropine eye drops in children with strabismus or after the strabismus surgery.

Strabismus is a common eye disease in children, with an incidence rate of about 3%. It is reported that about 72% of strabismus cases in Asia are exotropia, of which intermittent exotropia is the most common type, and most cases are accompanied with myopia. It is found that patients with intermittent exotropia are often associated with abnormal accommodation. Ha SG reported that the amount of accommodation required to maintain binocular fusion in patients with intermittent exotropia was greater than that of normal controls. In addition, pupil size and visual clarity are also factors affecting accommodation. In conclusion, atropine eye drops may affect the occurrence and development of intermittent exotropia by reducing the amplitude of accommodation, dilating pupils and blurred near vision. At the same time, the reduction of accommodation causes poor focusing and inappropriate afferent signals of the convergence system, which will lead to the fatigue of the convergence and divergence system, which may affect the ocular alignment of exotropia after surgery. In most cases, the reduced accommodation and convergence might induce exotropia, but in some patients, they may use more accommodative stimuli to compensate the insufficiency of accommodation, and there may be an increase in convergence or even esotropia.

In general, in China, myopia with exotropia or exophoria is a high incidence of eye disease in children, and low concentration atropine eye drops have been widely used to control the progression of myopia. It is urgent to carry out a large sample randomized controlled clinical trial to evaluate the impact of low concentration atropine on the ocular alignment and binocular vision of patients with exotropia and exophoria, and guide much safer application of the low concentration atropine eye drops.

ELIGIBILITY:
Inclusion Criteria:

* The age ranged from 5 to 14 years;
* Astigmatism < 2.5D, spherical power: - 1.00D ~ -6.00D; difference between eyes in spherical power < 1.5D, difference between eyes in astigmatism < 1.00D;
* Intraocular pressure < 21mmHg;
* Ocular alignment fulfilling the following criteria：Exophoria with an exodeviation at near > 6PD12; Intermittent exotropia with an exodeviation ≤25 PD both at distance and at near, Titmus <=400 arc seconds; Intermittent exotropia patients underwent strabismus surgery, 6 months after operation, fulling the criteria of exophoria and intermittent exotropia mentioned before.
* Subjects and their parents or legal guardians have signed informed consent and are willing to accept randomized grouping and regular follow-up.

Exclusion Criteria:

* Amblyopia
* Have heart disease or serious respiratory disease
* Allergic to atropine, cyclopentantone, propoxybenzocaine and benzalkonium chloride;
* Those who have used contact lenses, bifocal lenses, or other measures to control myopia (including atropine);
* No binocular vision;
* Combined with vertical strabismus≥5PD, abnormal oblique muscle function≥ 2+, cyclodeviation, DVD or A-V pattern, paralytic and restrictive strabismus, comitant esotropia；
* Previous history of other ocular surgery;
* Severe complications during or after strabismus surgery, such as perforation of the sclera, tear and detachment of extraocular muscle; postoperative eye movement limitation; visual acuity decreased after operation;
* Combined with other ocular diseases;
* Craniofacial malformations affecting the orbits;
* significant neurological disorders;
* Birth less than 34 weeks or birth weight less than 1500 g;
* Intraocular pressure > 21mmhg;
* Unable to cooperate with the examination.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 339 (Estimated)
Dates: Start 2024-03-02 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Refraction | 1 year and 2 years
  Change from baseline in spherical equivalent measured using cycloplegic autorefraction
Axial length | 1 year and 2 years
  Change from baseline in Axial length measured using Optical Biometer

SECONDARY OUTCOMES:
Stereopsis | 1 year and 2 years
  Change from baseline in stereopsis measured with the Random dot stereogram.
Fusion | 1 year and 2 years
  Change from baseline in fusion measured with the Worth Four-Dots.
AC/A ratio | 1 year and 2 years
  Change from baseline in AC/A ratio measured using the Von Graefe method
Negative and positive relative accommodation | 1 year and 2 years
  Change from baseline in negative and positive relative accommodation measured using a phoropter.
Fusional convergence and divergence amplitudes | 1 year and 2 years
  Change from baseline in fusional convergence and divergence amplitudes measured using a phoropter.
Accommodative facility | 1 year and 2 years
  Change from baseline in accommodative facility measured using flip lens technique.
Accommodative amplitude | 1 year and 2 years
  Change from baseline in accommodative amplitude measured using the minus lens techniques.
Near point of convergence | 1 year and 2 years
  Change from baseline in near point of convergence measured using standard push-up technique.
Ocular alignment | 1 year and 2 years
  Change from baseline in ocular alignment measured by a prism alternating cover test using an accommodative target at 6 m and 1/3 m.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye and ENT Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
The investigators concerns about patient privacy issues and it's better to protect the publication potential.

REFERENCES:
- [Background] Chia A, Chua WH, Cheung YB, Wong WL, Lingham A, Fong A, Tan D. Atropine for the treatment of childhood myopia: safety and efficacy of 0.5%, 0.1%, and 0.01% doses (Atropine for the Treatment of Myopia 2). Ophthalmology. 2012 Feb;119(2):347-54. doi: 10.1016/j.ophtha.2011.07.031. Epub 2011 Oct 2. PMID 21963266
- [Background] Chia A, Chua WH, Wen L, Fong A, Goon YY, Tan D. Atropine for the treatment of childhood myopia: changes after stopping atropine 0.01%, 0.1% and 0.5%. Am J Ophthalmol. 2014 Feb;157(2):451-457.e1. doi: 10.1016/j.ajo.2013.09.020. Epub 2013 Dec 4. PMID 24315293
- [Background] Yam JC, Jiang Y, Tang SM, Law AKP, Chan JJ, Wong E, Ko ST, Young AL, Tham CC, Chen LJ, Pang CP. Low-Concentration Atropine for Myopia Progression (LAMP) Study: A Randomized, Double-Blinded, Placebo-Controlled Trial of 0.05%, 0.025%, and 0.01% Atropine Eye Drops in Myopia Control. Ophthalmology. 2019 Jan;126(1):113-124. doi: 10.1016/j.ophtha.2018.05.029. Epub 2018 Jul 6. PMID 30514630
- [Background] Ha SG, Jang SM, Cho YA, Kim SH, Song JS, Suh YW. Clinical exhibition of increased accommodative loads for binocular fusion in patients with basic intermittent exotropia. BMC Ophthalmol. 2016 Jun 7;16:77. doi: 10.1186/s12886-016-0260-y. PMID 27266700
- [Background] Jampolsky A. Ocular divergence mechanisms. Trans Am Ophthalmol Soc. 1970;68:730-822. No abstract available. PMID 5524219
- [Background] Rutstein RP, Daum KM. Exotropia associated with defective accommodation. J Am Optom Assoc. 1987 Jul;58(7):548-54. PMID 3668152
- [Background] Schor C, Horner D. Adaptive disorders of accommodation and vergence in binocular dysfunction. Ophthalmic Physiol Opt. 1989 Jul;9(3):264-8. doi: 10.1111/j.1475-1313.1989.tb00904.x. PMID 2622666
- [Background] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Background] Chia A, Lu QS, Tan D. Five-Year Clinical Trial on Atropine for the Treatment of Myopia 2: Myopia Control with Atropine 0.01% Eyedrops. Ophthalmology. 2016 Feb;123(2):391-399. doi: 10.1016/j.ophtha.2015.07.004. Epub 2015 Aug 11. PMID 26271839
- [Background] Chia A, Roy L, Seenyen L. Comitant horizontal strabismus: an Asian perspective. Br J Ophthalmol. 2007 Oct;91(10):1337-40. doi: 10.1136/bjo.2007.116905. Epub 2007 May 2. PMID 17475715
- [Background] Chen X, Fu Z, Yu J, Ding H, Bai J, Chen J, Gong Y, Zhu H, Yu R, Liu H. Prevalence of amblyopia and strabismus in Eastern China: results from screening of preschool children aged 36-72 months. Br J Ophthalmol. 2016 Apr;100(4):515-9. doi: 10.1136/bjophthalmol-2015-306999. Epub 2015 Aug 10. PMID 26261229
- [Background] Chen AH, O'Leary DJ, Howell ER. Near visual function in young children. Part I: Near point of convergence. Part II: Amplitude of accommodation. Part III: Near heterophoria. Ophthalmic Physiol Opt. 2000 May;20(3):185-98. No abstract available. PMID 10897340
- [Background] Mohney BG, Holmes JM. An office-based scale for assessing control in intermittent exotropia. Strabismus. 2006 Sep;14(3):147-50. doi: 10.1080/09273970600894716. PMID 16950743